CLINICAL TRIAL: NCT03739515
Title: A Pilot Randomised Controlled Trial Exploring the Impact of a Dedicated Health and Social Care Professionals (HSCP) Team in the Emergency Department on the Quality, Safety and Cost-effectiveness of Care for Older Adults
Brief Title: Impact of an Allied Health Team in the Emergency Department on Older Adults' Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Limerick (Other)
Collaborators: University Hospital of Limerick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Optimend_WP4
Record Dates: First submitted 2018-11-07; First posted 2018-11-13 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: ED-based Allied Health Services
Keywords: Emergency department; Health and Social Care Professional; Team care; Older patients; Effectiveness
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly assigned to either the experimental group (ED-based HSCP intervention) or the control group (ED routine care). By assigning participants at random, it is possible to infer that any observed group differences are attributable to the independent variable (the intervention under investigation).
Who Masked: Outcomes Assessor
Masking Description: To minimise the possibility of selection bias, a person independent of the recruitment process will complete random group allocation. Computer generated random numbers will be created and placed in sealed envelopes by this independent person. These numbers will be stored in the pre-sealed envelopes in a locked drawer in the Health Research Institute at the Clinical Education and Research Centre (CERC). Allocation will be revealed after recruitment by a telephone call from the dedicated research nurse to this independent person, who will open the next envelope in the sequence and give the randomisation information to the research nurse. Each envelope will be opened on enrolment of an eligible participant. After allocation is revealed, the appropriate intervention will be organised by the team.
  In addition, the outcome assessment will be conducted by a research nurse blinded to the patient allocation in order to reduce potential detection bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSCP team (Experimental): Patients in this arm will receive comprehensive assessment and/or pre-discharge services by an ED-based HSCP team
  Interventions: Other: HSCP intervention
- Routine care (Active Comparator): Patients in this arm will receive routine ED care
  Interventions: Other: ED routine care

INTERVENTIONS:
Other: HSCP intervention — A team of HSCPs (physiotherapist, occupational therapist, medical social worker) will provide comprehensive functional assessment to older patients
  Arms: HSCP team
Other: ED routine care — ED staff including consultants and nurses will provide patients with routine ED medical care.
  Arms: Routine care

SUMMARY:
The study aims to examine the impact of implementing a dedicated team of Health and Social Care Professionals (HSCPs) in the emergency department (ED) of a large Irish hospital on the quality, safety and cost-effectiveness of care for older adults (aged ≥65). Early assessment and intervention provided by the HSCP team will be compared to routine ED care to explore potential benefits related to key ED outcomes, including length of stay as well as hospital admissions and patient satisfaction/quality of life.

This study is part of an ongoing interdisciplinary project funded by the Health Research Board of Ireland through the Research Collaborative on Quality and Patient Safety (RCQPS) Grant Call 2017. The project is led by Dr Rose Galvin, Senior Lecturer in Physiotherapy at the University of Limerick (UL, Ireland), and overseen by an interdisciplinary steering group of expert researchers and clinicians in Emergency Medicine and Allied Health.

DETAILED DESCRIPTION:
Background Internationally, emergency departments (EDs) face significant challenges in delivering high quality and timely patient care on an ever-present background of increasing patient numbers and limited hospital resources. Research demonstrates that ED crowding contributes to a reduction in the quality of patient care, delays in commencement of treatment and that adherence with recognised clinical guidelines worsens [1].

Identifying quality improvement strategies to improve patient flow in the ED can enhance quality of care. Evidence from international studies demonstrates that Health and Social Care Professionals (HSCPs) such as physiotherapists, occupational therapists and medical social workers can play a role in the ED in reducing length of patient stay, avoiding unnecessary hospital admissions and improving patient experience [2,3]. However, the quality of the evidence is mixed, primarily due to weaknesses in designing the studies.

Aim The overall aim of the study is to examine the impact of a dedicated team of Health and Social Care Professionals (HSCPs) in the Emergency Department (ED) on the quality, safety and cost-effectiveness of care of older adults in the ED.

The objectives of the study are as follows:

1. To implement a HSCP team including a whole time equivalent senior physiotherapist (PT), senior occupational therapist (OT) and senior medical social worker (MSW) in the Emergency Department at University Hospital Limerick (UHL) for a period of six months.
2. To examine if early assessment and intervention by the HSCP team improves the quality, safety and cost-effectiveness of care among older adults who present to the ED, as compared to usual care.
3. To conduct a process evaluation of the HSCP intervention through focus group interviews with the HSCP team and representation from the wider ED staff regarding the implementation, delivery and impact of the intervention.

Methods

Study design The study represents a pilot randomised controlled trial which will compare assessment and/or interventions carried by a HSCP team, comprised of a physiotherapist, an occupational therapist and a medical social worker, in the ED with usual ED care. The Consolidated Standards of Reporting Trials (CONSORT) reporting guidelines will be followed to ensure the standardised conduct and reporting of the research.

Population All adults ≥65 years who present to the Emergency Department at University Hospital Limerick (UHL) between December 2018 and March 2019 (inclusive) will be considered eligible for inclusion to the study provided that they meet the inclusion criteria (see below). However, similar to other studies, the HSCP team is operational between the hours of 8am and 5pm Monday-Friday. Therefore, individuals who present outside of these hours may not be offered/included in the study.

Consent Potential participants will initially be informed of the study by the triage nurse or the treating physician. If participants indicate a willingness to hear more about the study, the dedicated research nurse on the project will be informed. The research nurse will subsequently meet with the potential participant and describe the study in detail and provide potential participants with an information leaflet. Participants will be given the opportunity to ask further questions about the project should they wish to do so. Written informed consent will be obtained by the research nurse if/when the participant indicates their willingness to formally participate in the study. Participants will have the duration of their index admission to consider participation in the study. Consent and mechanisms relating to data controlling and processing will be compliant with the European Union (EU) General Data Protection Regulation (GDPR) 2016/679 and also in compliance with the Data Protection Act 2018 [(Section 36(2)) (Health Research) Regulations 2018].

Intervention The intervention will comprise initially of a detailed assessment by one or more members of the dedicated HSCP team (physiotherapy, occupational therapy and medical social work). The assessment will include but not be limited to an assessment of mobility and stairs, transfer, personal care, activities of daily living (ADLs), social supports, cognition, lying & standing blood pressures. Members of the HSCP team will be guided by their clinical expertise and codes of professional practice. Similarly, interventions prescribed by the HSCP team will be based on subjective and objective assessment of patients and will include mobility aids, exercise programmes, ADL equipment and onward referral as appropriate. All assessments and interventions will be included in the medical chart of individual participants.

Comparison The comparison group will receive routine care for the duration of their stay in the ED. Currently there is no dedicated team of HSCPs in the Emergency Department at UHL. Ad-hoc services are provided by allied health professionals if they are requested by a member of the team in the ED. This process will continue for the duration of the trial.

Outcomes and analysis The primary outcome of the study is duration of patient ED stay (mean hours from time of arrival to discharge or admission). Secondary outcomes will include the incidence of inpatient admission from the ED (defined as the proportion of patients who are admitted to hospital after their index visits), the duration of hospital admission after the ED index visit, as well as the number of ED re-attendances, nursing home admissions, unplanned hospital visits (and duration of stay) and mortality within 30 days, four months and six months of the initial index visit. Healthcare utilisation (visits to GP, public health nurse, home help, private consultations, outpatient department visits, or allied health services) will also be captured at 30 days, four months and six months. Assessment of patient oriented outcomes include the Barthel Index for Activities of Daily Living (17) as a global measure of function and the EuroQoL's 5-Dimension 5-Level (EQ-5D-5L) to measure health-related quality of life (18), which will be conducted at baseline as well as at follow-up (30 days and six months, with quality of life also assessed at four months).

In addition, patient satisfaction with their index visit will be explored using the 18-item Patient Satisfaction Questionnaire (PSQ-18) (19) at the time of the visit.

An economic analysis will estimate the incremental cost effectiveness of the HSCP team from the perspective of the Irish public health service, as compared to usual care. We will estimate health care costs from reference costs from national data sources. Participants' responses to the EQ-5D-5L questionnaire will be used to estimate health states utilities using the Irish value set (20) and Quality-Adjusted Life Years (QALYs) for each treatment group will be estimated across all timepoints.

Lastly, a process evaluation will be conducted through a mixed quantitative-qualitative design to describe the implementation of the intervention as well as investigate the mechanisms and contextual influences of the implementation as perceived by the HSCP team and representation from the wider ED staff. A detailed study protocol for the process evaluation is in preparation.

Each participant in the study will be assigned a numerical code in order to link data collected at baseline to the data collected at follow-up at 30 days, four and six months. Aggregate data will be anonymised. Appropriate descriptive statistics will be used to describe the baseline characteristics of study participants. These will include proportions, percentages, ranges, means and standard deviations and medians and interquartile ranges (where data are not normally distributed). We will analyse differences across the two groups for all continuous outcomes (ED length of stay, etc.) by using independent samples t-tests with 95% CI. The non-parametric equivalent will be used for skewed data. Incidence of ED return, unplanned hospital admission, nursing home admission and healthcare utilization will be explored using crude and adjusted risk ratios with associated 95% Confidence Interval (CI).

Considering the cost-effectiveness analysis, as per the Irish Health Information and Quality Authority (HIQA) guidance (21), the primary endpoint of the cost-effectiveness analysis will be costs, QALYs and the Incremental Cost Effectiveness Ratio (ICER). Analysis of uncertainty of the joint distribution of cost and QALYs between the two arms of the study will be presented on a cost-effectiveness acceptability curve to indicate the probability that the HSCP intervention will be cost effective, based on available trial data and across various willingness to pay thresholds.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years
* Medically stable (treating physician)
* Off baseline mobility
* Capacity (Mini Mental State Examination score ≥17) and willingness to provide informed consent
* Presenting during HSCP operational hours (8am-5pm Monday-Friday)

Exclusion Criteria:

* Under 65 years
* Medically unstable
* Neither the patient nor the carer can communicate in English sufficiently to complete consent or baseline assessment
* Present outside HSCP operational hours.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 354 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
ED length of stay | 1-24 hours (one day) after accessing the ED
  Hours from ED admission to discharge

SECONDARY OUTCOMES:
Incidence of Representations | 30 days, four months, and six months after index visit
  Percentages of patients who experience ED revisits, unplanned hospital visits or nursing home admissions after the ED index visit
Incidence of Healthcare utilization | 30 days, four months, and six months after index visit
  Percentages of patients who visit a general practitioner (GP), a public health nurse, outpatient departments, private consultations, home help, or allied health services after the ED index visit
Functional status | Baseline, 30 days and six months after index visit
  Patient global functioning as measured through the Barthel Index of Activities of Daily Living.
  The Barthel Index is a 10-item scale used to assess functional independence. The scoring varies across items:
  * bowels, bladder, toilet use, feeding, dressing, and stairs are scored from from 0 (dependence or inability) to 2 (independence)
  * grooming and bathing are scored either 0 (dependent or needs help) or 1 (independent)
  * transfer and mobility are scored 0 (dependent), 1 (major help), 2 (minor help), or 3 (independent).
  The total score ranges from 0 to 20 and it is obtained by adding up the scores of each item. Lower scores indicated increased disability. In case of rehabilitation, changes of more than two points in the total score reflect a probable genuine change, and change on one item from fully dependent to independent is also likely to be reliable.
Patient quality of life | Baseline, 30 days, four months and six months after index visit
  Quality of life assessed through the EuroQoL-5D-5L (EQ-5D-5L). The EQ-5D-5L is a standardised instrument developed by the EuroQoL Group (https://euroqol.org/euroqol/) to measure health-related quality of life.
  It includes a descriptive questionnaire assessing 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) with 5 levels of self-rated severity (1 = no problems, 2 = slight problems, 3 = moderate problems, 4 = severe problems, and 5 = extreme problems). Each dimension is scored separately from 0 to 5 and the patient's "health state" is coded as a 5-digit string.
  It also includes a vertical visual analogue scale (VAS) to record the patient's self-rated health on a scale from 0 (worst health) to 100 (best health). The score assigned by the patient represents the self-reported level of health.
Patient satisfaction with index visit | At time of index visit
  Patient satisfaction with the index visit will be assessed using the Patient Satisfaction Questionnaire (PSQ-18) - Short Form.
  The PSQ-18 is an 18-item questionnaire that assesses patient's satisfaction with 6 aspects of care: technical quality, interpersonal manner, communication, financial aspects, time spent with the healthcare provider, and accessibility of care. General satisfaction is also assessed.
  The items are presented as statements about the experience of care and rated based on the patient's level of agreement with each statement from 1 (strongly agree) to 5 (strongly disagree).
  The PSQ-18 yields separate scores for each of seven different dimensions. All items should be scored so that high scores reflect satisfaction with medical care. After item scoring, items within the same sub-scale should be averaged together to create the 7 sub-scale scores.
Process evaluation | Within two months after completion of data collection (eight months after beginning of the study)
  The level of staff satisfaction and their perceptions on the implementation, delivery and impact of the intervention will be assessed with the HSCP team and other ED staff members (consultants, nurses) using qualitative methodologies (focus groups) after the completion of participant recruitment.
Cost-effectiveness | Four months after index visit
  An economic analysis will estimate the incremental cost effectiveness of the HSCP team from the perspective of the Irish public health service, as compared to usual care. We will estimate health care costs from reference costs from national data sources. Participants' responses to the EQ-5D-5L questionnaire will be used to estimate health states utilities using the Irish value set (20) and Quality-Adjusted Life Years (QALYs) for each treatment group will be estimated across all timepoints
Nursing home admission | 30 days and six months after index visit
  The rates of patients admitted to a nursing home will be captured at follow-up
Mortality | 30 days and six months after the index visit
  The rates of patients deceased will be captured at follow-up
Hospital admission rate | Within 72 hours of ED index visit
  Percentages of patients admitted to the ward from the ED

CONTACTS AND LOCATIONS:
Overall Officials: Rose Galvin, PhD, Principal Investigator — University of Limerick; Damien Ryan, PhD, Principal Investigator — University Hospital of Limerick
Locations (1):
- University Hospital Limerick, Limerick, Co. Limerick, Ireland

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers

REFERENCES:
- [Background] Carter EJ, Pouch SM, Larson EL. The relationship between emergency department crowding and patient outcomes: a systematic review. J Nurs Scholarsh. 2014 Mar;46(2):106-15. doi: 10.1111/jnu.12055. Epub 2013 Dec 19. PMID 24354886
- [Background] Arendts G, Fitzhardinge S, Pronk K, Hutton M. Outcomes in older patients requiring comprehensive allied health care prior to discharge from the emergency department. Emerg Med Australas. 2013 Apr;25(2):127-31. doi: 10.1111/1742-6723.12049. Epub 2013 Feb 19. PMID 23560962
- [Background] Cassarino M, Robinson K, Quinn R, Naddy B, O'Regan A, Ryan D, Boland F, Ward ME, McNamara R, McCarthy G, Galvin R. Effectiveness of early assessment and intervention by interdisciplinary teams including health and social care professionals in the emergency department: protocol for a systematic review. BMJ Open. 2018 Jul 16;8(7):e023464. doi: 10.1136/bmjopen-2018-023464. PMID 30012796
- [Derived] Trepel D, Ruiz-Adame M, Cassarino M, Ahern E, Devlin C, Robinson K, O'Shaughnessy I, McCarthy G, Corcoran C, Galvin R. The cost effectiveness of early assessment and intervention by a dedicated health and social care professional team for older adults in the emergency department compared to treatment-as-usual: Economic evaluation of the OPTI-MEND trial. PLoS One. 2024 Jun 25;19(6):e0298162. doi: 10.1371/journal.pone.0298162. eCollection 2024. PMID 38917081
- [Derived] Cassarino M, Cronin U, Robinson K, Quinn R, Boland F, Ward ME, McNamara R, O'Connor M, McCarthy G, Ryan D, Galvin R. Development and delivery of an allied health team intervention for older adults in the emergency department: A process evaluation. PLoS One. 2022 May 26;17(5):e0269117. doi: 10.1371/journal.pone.0269117. eCollection 2022. PMID 35617330
- [Derived] Cassarino M, Robinson K, Trepel D, O'Shaughnessy I, Smalle E, White S, Devlin C, Quinn R, Boland F, Ward ME, McNamara R, Steed F, O'Connor M, O'Regan A, McCarthy G, Ryan D, Galvin R. Impact of assessment and intervention by a health and social care professional team in the emergency department on the quality, safety, and clinical effectiveness of care for older adults: A randomised controlled trial. PLoS Med. 2021 Jul 28;18(7):e1003711. doi: 10.1371/journal.pmed.1003711. eCollection 2021 Jul. PMID 34319971
- [Derived] Griffin A, O'Neill A, O'Connor M, Ryan D, Tierney A, Galvin R. The prevalence of malnutrition and impact on patient outcomes among older adults presenting at an Irish emergency department: a secondary analysis of the OPTI-MEND trial. BMC Geriatr. 2020 Nov 7;20(1):455. doi: 10.1186/s12877-020-01852-w. PMID 33160319
- [Derived] Cassarino M, Robinson K, O'Shaughnessy I, Smalle E, White S, Devlin C, Quinn R, Trepel D, Boland F, Ward ME, McNamara R, O'Connor M, McCarthy G, Ryan D, Galvin R. A randomised controlled trial exploring the impact of a dedicated health and social care professionals team in the emergency department on the quality, safety, clinical and cost-effectiveness of care for older adults: a study protocol. Trials. 2019 Oct 15;20(1):591. doi: 10.1186/s13063-019-3697-5. PMID 31615573
- [Derived] Cassarino M, Cronin U, Robinson K, Quinn R, Boland F, Ward ME, MacNamara R, O'Connor M, McCarthy G, Ryan D, Galvin R. Implementing an allied health team intervention to improve the care of older adults in the emergency department: protocol for a process evaluation. BMJ Open. 2019 Jul 16;9(7):e032645. doi: 10.1136/bmjopen-2019-032645. PMID 31315881